CLINICAL TRIAL: NCT04224363
Title: Whether it is More Appropriate to Spray Lugol's Solution From Cervical Esophagus to Esophagogastric Junction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2020SDU-QILU-G001
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Lugol's solution; staining sequence; Esophageal Squamous Cell Carcinoma; Effectiveness; Safety
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Downward Staining (Experimental): This group patients were given Lugol's solution staining from cervical esophagus to esophagogastric junction （downward）during chromemdoscopy.
  Interventions: Procedure: staining from cervical esophagus to esophagogastric junction
- Upward Staining (Experimental): This group patients were given Lugol's solution staining from esophagogastric junction to cervical esophagus（upward）during chromemdoscopy.
  Interventions: Procedure: staining from esophagogastric junction to cervical esophagus

INTERVENTIONS:
Procedure: staining from cervical esophagus to esophagogastric junction — This group patients were given Lugol's solution staining from cervical esophagus to esophagogastric junction （downward）during chromemdoscopy.
  Arms: Downward Staining
Procedure: staining from esophagogastric junction to cervical esophagus — This group patients were given Lugol's solution staining from esophagogastric junction to cervical esophagus（upward）during chromemdoscopy.
  Arms: Upward Staining

SUMMARY:
The aim of this study is to compare the effectiveness and safety of spraying Lugol's solution from cervical esophagus to esophagogastric junction (downward) and from esophagogastric junction to cervical esophagus （upward）during chromoendoscopy.

DETAILED DESCRIPTION:
Chromoendoscopy using Lugol's solution is effective for the detection of early esophageal squamous neoplasia. However, there is no study to investigate the sequence of Lugol's staining during endoscopic procedure.

The aim of this study is to compare the effectiveness and safety of spraying Lugol's solution from cervical esophagus to esophagogastric junction (downward) and from esophagogastric junction to cervical esophagus （upward）during chromoendoscopy.

ELIGIBILITY:
Inclusion Criteria:

* High risk patients of early esophageal squamous neoplasias.

Exclusion Criteria:

* After esophageal surgery or endoscopic treatment ;
* Known esophageal radiotherapy or chemotherapy ;
* Esophageal stenosis;
* Acute bleeding;
* A known allergy to iodine;
* Coagulopathy (prothrombin time <50% of control, partial thromboplastin time >50 seconds);
* Having food retention;
* Severe hepatic ,renal, cardiovascular or metabolic dysfunction ;
* Being pregnant or lactating.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Image Quality | intraoperative
  Image quality is blindly quantified by a 4-point scale from the endoscopists. A higher score representing higher image quality.

SECONDARY OUTCOMES:
Adverse events | 24 hours
  Adverse events of the two groups.
Dose | intraoperative
  Usage of Lugol's solution in each group.
Effectiveness | 1 month
  Detection rate of esophageal squamous cell carcinoma of the two groups.
Tolerance | intraoperative
  The 4-point scale was used to assess the tolerance of endoscopist to the esophageal spasm caused by Lugol's solution which prevent endoscopy from passing. 1-4 means the resistance as intolerable, tolerable, mild, or non-existing.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, MD,PhD, Principal Investigator — Qilu Hospital of Shandong University